CLINICAL TRIAL: NCT04885205
Title: Use of Cognitive Behavioral Therapy for Insomnia in Individuals With a Concussion
Brief Title: Use of CBT-I in Individuals With a Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00146439
Record Dates: First submitted 2021-03-09; First posted 2021-05-13 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Concussion, Mild
MeSH Terms: conditions — Brain Concussion | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I Initial Group (Experimental): The CBT-I Initial Group will start the CBT-I intervention immediately following baseline assessments. After re-assessment 1, participants in the CBT-I Initial Group will continue with typical activities while the WL group will receive the CBT-I intervention. After re-assessment 2, both groups continue typical activities. All participants will complete a third re-assessment 21 weeks after starting the study.
  Interventions: Behavioral: cognitive behavioral therapy for insomnia (CBT-I)
- Wait List Group (Active Comparator): The WL will wait 6 weeks before starting the CBT-I intervention. After re-assessment 1, participants in the CBT-I Initial Group will continue with typical activities while the WL group will receive the CBT-I intervention. After re-assessment 2, both groups continue typical activities. All participants will complete a third re-assessment 21 weeks after starting the study.
  Interventions: Behavioral: cognitive behavioral therapy for insomnia (CBT-I)

INTERVENTIONS:
Behavioral: cognitive behavioral therapy for insomnia (CBT-I) — The CBT-I program is a 6-week, 1x/week, one-on-one program. The delivery of CBT-I will be done remotely over a secure teleconference service (Zoom) or phone. Participants will maintain a sleep diary during the course of the program to aid in tailoring the intervention. Each session lasts about 45-60min:

SUMMARY:
Sleep disturbances have been shown to contribute to poorer recovery from a concussion. Furthermore, sleep disturbances have been associated with more frequent and severe post-concussion symptoms including headache, vertigo, anxiety, depression, and decreased short term memory reducing quality of life and productivity at work or school. Additionally, recent research indicates that individuals with a concussion who have poor sleep quality have increased levels of Neurofilament light (NfL) and tau biomarkers indicating that there may still be axonal damage after weeks or months after the initial concussion injury. Post-concussion symptoms have been associated with higher levels of these biomarkers and there has been a report of higher levels of NfL and tau years following a concussion event. Cognitive behavioral therapy for insomnia (CBT-I) is an effective treatment for insomnia yet it remains unclear if this treatment method is effective in improving sleep outcomes, reducing concomitant post-concussion symptoms, and biomarkers of neural injury/risk in individuals post- concussion. The central hypothesis for this project is treating sleep disturbances will yield a clinically relevant reduction in concomitant post-concussion symptoms. The objective for the proposed study is to determine if CBT-I will reduce insomnia symptoms and improve concomitant post-concussion symptoms in individuals after concussion and if symptom improvements are maintained at 6-weeks and 12-weeks after CBT-I intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 64 years old
* At least 4 weeks since concussion injury
* Self-report difficulty falling asleep, maintaining sleep, or waking up too early at least 3 nights per week since injury
* Score ≥10 on the Insomnia Severity Index to indicate clinical insomnia.
* Score ≥25 on the Mini-Mental State Examination (MMSE) questionnaire

Exclusion Criteria:

* Known untreated sleep disorder (such as sleep apnea, restless leg syndrome, circadian rhythm disorder, hypersomnia, parasomnias)
* Increased risk obstructive sleep apnea (STOP BANG Score ≥3)
* Increased risk of restless leg syndrome on RLS-Diagnosis Index
* Increased risk of circadian rhythm sleep-wake disorder (respond "Yes" to all circadian rhythm questions).
* Increased risk of parasomnia (Respond "Yes" to all questions for night mere disorder OR respond "Yes" to all REM sleep arousal disorder: Sleep walking questions, OR responds " Yes" to all REM sleep arousal disorder: Sleep Terrors questions, OR respond "Yes" to all REM sleep behavior disorder questions.)
* Active abuse or history (up to 2 years) of alcohol/ drug dependence as defined by the DSM-V criteria
* Severe mental illness such as schizophrenia or bipolar disorder
* Score of > 29 on the Beck Depression Inventory or indication of suicidality (response of "2" or "3"to item 9)
* History of diagnosed nervous system disorder other than concussion (such as multiple sclerosis, Parkinson's Disease, Stroke)
* Currently works nightshift

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
change in Insomnia Severity Index | baseline to 21 weeks
  7 questions each rated on a 0-4 scale. The range of scores on the ISI is 0-28
change in PSQI | baseline to 21 weeks
  Scores range from 0-21 with a higher score indicating a lower quality of sleep
change in Post-Concussion Symptom Scale | baseline to 21 weeks
  Severity of 22 concussion-related symptoms are assessed by a Likert scale 0-6. Participants will rate their symptoms from a "0" or no symptom to "6" extreme symptom. A score of 132 is the maximum someone can have indicating all symptoms are severe. 2. The number of post-concussion symptoms will be assessed by counting the number of symptoms that the participant identified as having a severity of "1" or higher on the PCSS. A score of a "1" indicates that the symptom is mild, but still noticeable.
change in Beck Anxiety Inventory | baseline to 21 weeks
  The tool consists of 21 items that are scored on a Likert scale of 1-3. Scores range from minimal anxiety (0-7), mild anxiety (8-15) moderate anxiety (16-25) and severe anxiety (<30).
change in Beck Depression Inventory | baseline to 21 weeks
  21 item questionnaire used to assess the severity of depression. Scores range from 1 to greater than 40.

SECONDARY OUTCOMES:
change in Dysfunctional Beliefs About Sleep (DBAS) | baseline to 21 weeks
  30 item Likert-scale self-report questionnaire with 0 = "strongly disagree" to 10 = "strongly agree"; scores range from 0-300 and a higher score indicates more dysfunctional beliefs about sleep
change in Sleep Self-Efficacy | baseline to 21 weeks
  9 item self-report Likert-scale questionnaire; Scores range from 0-45 and a higher score indicates higher sleep self-efficacy
change in RU-SATED questionnaire | baseline to 21 weeks
  to 6 questions asking sleep regularity, subjective satisfaction, appropriate timing, adequate duration, high sleep efficiency, and sustained alertness during the day; Participants answer each question with "Rarely/ Never" (0), " Sometimes" (1), and "Usually/ Always" (2). There are ten points possible.
change in plasma neurofilament light (NfL) | baseline to 21 weeks
  blood marker of axonal damage
change in plasma pTau181 | baseline to 21 weeks
  blood marker of tauopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Catherine Siengsukon, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ludwig R, Rippee M, D'Silva L, Radel J, Eakman AM, Morris J, Beltramo A, Drerup M, Siengsukon C. The Impact of Cognitive Behavioral Therapy for Insomnia on Neurofilament Light and Phosphorylated Tau in Individuals with a Concussion. Arch Clin Neuropsychol. 2025 Apr 27;40(3):437-444. doi: 10.1093/arclin/acae096. PMID 39504933
- [Derived] Ludwig R, Rippee M, D'Silva LJ, Radel J, Eakman AM, Morris J, Drerup M, Siengsukon C. Assessing Cognitive Behavioral Therapy for Insomnia to Improve Sleep Outcomes in Individuals With a Concussion: Protocol for a Delayed Randomized Controlled Trial. JMIR Res Protoc. 2022 Sep 23;11(9):e38608. doi: 10.2196/38608. PMID 36149737